CLINICAL TRIAL: NCT01678508
Title: Pharmacogenetically Based Dosing of Thiopurines in Childhood Acute Lymphoblastic Leukemia - Influence on Cure Rates and Risk of Second Cancer
Brief Title: Pharmacogenetically Based Dosing of Thiopurines in Childhood Acute Lymphoblastic Leukemia
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Kjeld Schmiegelow, Professor MD, Rigshospitalet, Denmark
Other Study IDs: NOPHO ALL2000 TPMT and outcome
Record Dates: First submitted 2012-05-22; First posted 2012-09-05 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-09

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — whole blood stored for a subset of patients
Oversight: Data Monitoring Committee: No

SUMMARY:
In a population-based study to explore the impact of TPMT-status on the risk of relapse and of second cancer among all patients treated according to the NOPHO ALL2000.

DETAILED DESCRIPTION:
The thiopurines 6-mercaptopurine (6MP) and 6-thioguanine (6TG) are widely used in the treatment of childhood acute lymphoblastic leukemia (ALL). They primarily exert their cytotoxicity through conversion into 6-thioguanine nucleotides (6TGN) that are incorporated into DNA. Interindividual variations in response to thiopurine therapy are influenced by genetically determined polymorphisms in the activity of the enzyme thiopurine methyltransferase (TPMT). TPMT competes with the formation of 6TGN, as it methylates the thiopurines (especially 6MP) and some of their metabolites. Approximately ten percent of all individuals are TPMT heterozygous, with one wild type and one low activity allele, and one in three hundred individuals are TPMT deficient with two low activity alleles. During the maintenance therapy phase of the treatment of childhood ALL, which may last several years, 6MP is given on a daily basis at a starting dose of 75 mg/m.sq./day, which is subsequently adjusted to a white blood cell count of 1.5-3.5 x109/L. We have previously demonstrated that the risk of relapse is reduced by more than 50%, but the risk of second cancer was increased 3-fold among TPMT low activity patients. Accordingly, the Nordic ALL2000 protocol recommended the dosing of 6MP to be based on the patients TPMT activity. In the present study of almost 1000 Nordic patients, we will explore whether this strategy of TPMT-based individualised 6MP dosing have benefitted the patients by reducing their risk of second cancer while preserving their low risk of relapse.

ELIGIBILITY:
Inclusion Criteria:

* included in the NOPHO ALL2000 protocol
* entered 6-mercaptopurine/Methotrexate maintenance therapy in first remission
* available TPMT phenotype and/or genotype

Exclusion Criteria:

* children with Down Syndrome

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study cohort is based on patients enrolled in the NOPHO ALL2000 protocol.
Sampling Method: Probability Sample
Enrollment: 1020 (Actual)
Dates: Start 2002-01; Primary Completion 2011-07 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Cumulative risk of relapse and risk of second cancer by Kaplan-Meier analysis with Gray's test comparisons at 10 years | Up to 10 years from diagnosis
  The risks will be reported as percentages.

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Schmiegelow, M.D., Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark